CLINICAL TRIAL: NCT04538326
Title: Exercise Intensity During Interactive Video Games and Standard of Care of Individuals Post-Stroke
Brief Title: Exercise Intensity and Video Games: Persons Post-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Judith E Deutsch, PT, PhD, Professor and Director Rivers Lab, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro20160000916
Record Dates: First submitted 2020-04-07; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Stroke
Keywords: active video games; virtual reality; exercise intensity; Parkinson Disease
MeSH Terms: conditions — Stroke; Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Repeated measures, counter-balanced
Masking Description: Participants were told that the purpose of the study was to learn more about what type of exercise they liked. There was no indication that intensity was an outcome measure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single (Other): Participants exercised in two counter balanced blocks: repeated (standard of care and self-paced repeated custom game) and random (Kinect game and game-paced random custom game). Exercise bouts were for 8.5 minutes with ten minutes of rest in between so they could return to physiological baseline. Data were collected in a single session lasting two hours.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Participants performed stepping movements that were either cued by the investigator or interacted with a video game. There were three video game exercises that all involved stepping in either a repeated or a random pattern that was either self-paced or game paced.
  Other Names: Video Game Play; Standard of Care Stepping Activities

SUMMARY:
Persons post stroke executed stepping activities under four conditions: standard of care, interacting with: an off-the-shelf Microsoft-Kinect game, with a self-paced repeated custom video game and a game-paced random custom video game. Exercise intensity (neuromuscular and cardiovascular), enjoyment and perceived effort were measured during and after each condition.

DETAILED DESCRIPTION:
Persons post stroke were first familiarized with the four exercise conditions and then instrumented with a metabolic system and heart rate sensor. They played the games in two counter balanced blocks: repeated (standard of care and self-paced repeated custom) and random (Microsoft-Kinect game and game-paced random custom). Games were played for 8.5 minutes with ten minutes of rest in between so they could return to physiological baseline. During exercise they reported exertion and at the end of teach exercise trial they completed an enjoyment questionnaire. At the end of the first block, participants removed the metabolic system's mask and were assessed for motor recovery. Performances were video taped. At the end of data collection preferences for the activities were ranked and participants answered open ended questions. Data for neuromuscular and cardiovascular intensity, enjoyment and perceived effort were reduced and analyzed using a Repeated Measures Analysis of Variance (RMANOVA) with the appropriate post-hoc corrections. Where possible clinically meaningful changes were calculated.

ELIGIBILITY:
Inclusion Criteria:

* men and women post-stroke at least six months T
* able to ambulate 100 feet without physical assistance but allowed to use assistive devices and orthotics,
* able to stand for 3 minutes.
* cleared for exercise with the PARQ.

Exclusion Criteria:

1. history of severe heart disease, heart attack, valve replacement or coronary artery bypass surgery, severe lung disease, uncontrolled diabetes, traumatic brain injury or neurological disorder other than stroke
2. Are unable to follow directions.
3. Do not have adequate vision and hearing ability (either aided or unaided with glasses, contacts or hearing aids
4. Are unable to sign a consent form.
5. Unstable medical condition or musculoskeletal disorder such as severe arthritis, knee surgery, hip surgery, or any other condition that the investigators determine would impair the ability to perform the required stepping for the games presented.
6. Any other medical condition contraindications to exercise.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Neuromuscular intensity | collected continuously during each of the four conditions. Collected in a single 2 hour session
  movement repetitions (stepping and marching) measured through video tape measured continuously during each exercise bout
Cardiovascular intensity (metabolic Units) | collected continuously during each of the four conditions. Collected in a single 2 hour session
  metabolic units measured continuously during each exercise bout
Cardiovascular intensity (Percent of maximum heart rate) | collected continuously during each of the four conditions. Collected in a single 2 hour session
  the percent of the maximum heart rate
Enjoyment | four times collected in a single 2 hour session (once at the completion of each the four conditions).
  measured with the PACES questionnaire after each exercise bout
Borg Rate if Perceived Exertion Scale | Collected three times (at the beginning, middle and end) of each of the four exercise bouts during a single two hour session
  Measures perception of effort on a scale of 6-20

SECONDARY OUTCOMES:
Preference ranking | collected once at the end of the completed data collection of a 2 hour session
  ranking exercise preference from highest (1) to lowest (4)
Fugl Meyer Motor Assessment Scale_ Lower Extremity Section | collected once during the single 2 hour data collection session
  measure of lower extremity motor recovery

OTHER OUTCOMES:
Open ended questions | collected once during a single 2 hour data collection session
  questions about preference and exertion and anything else the participants wants to share

CONTACTS AND LOCATIONS:
Overall Officials: Judith Deutsch, PT, PhD, Principal Investigator — Rutgers University
Locations (1):
- School of Health Professions, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie the results of a publication will be available through the publishers repository. We
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available through the appropriate journal data sharing plan.
Access Criteria: For systematic reviews or other secondary analyses.

REFERENCES:
- [Result] Kafri M, Myslinski MJ, Gade VK, Deutsch JE. Energy expenditure and exercise intensity of interactive video gaming in individuals poststroke. Neurorehabil Neural Repair. 2014 Jan;28(1):56-65. doi: 10.1177/1545968313497100. Epub 2013 Jul 29. PMID 23897906
- [Result] Kafri M, Myslinski MJ, Gade VK, Deutsch JE. High metabolic cost and low energy expenditure for typical motor activities among individuals in the chronic phase after stroke. J Neurol Phys Ther. 2014 Oct;38(4):226-32. doi: 10.1097/NPT.0000000000000053. PMID 25198864
- [Derived] Deutsch JE, James-Palmer A, Damodaran H, Puh U. Comparison of neuromuscular and cardiovascular exercise intensity and enjoyment between standard of care, off-the-shelf and custom active video games for promotion of physical activity of persons post-stroke. J Neuroeng Rehabil. 2021 Apr 14;18(1):63. doi: 10.1186/s12984-021-00850-2. PMID 33853608

DOCUMENTS (2):
  • Informed Consent Form (2019-04-21): https://cdn.clinicaltrials.gov/large-docs/26/NCT04538326/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-04-21): https://cdn.clinicaltrials.gov/large-docs/26/NCT04538326/Prot_SAP_001.pdf